CLINICAL TRIAL: NCT03206333
Title: Automated Quantification of Coronary Artery Calcifications on Radiotherapy Planning CTs for Cardiovascular Risk Prediction in Breast Cancer Patients: the BRAGATSTON Study
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Erasmus Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Dr., UMC Utrecht
Other Study IDs: 16/721 (IRB UMC Utrecht)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Cardiovascular Diseases
Keywords: Breast cancer; Cardiovascular diseases; Coronary artery calcium; Prediction; Risk stratification; Deep learning technique; Software development; Computed tomography scan
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients treated with radiotherapy

SUMMARY:
The aim of the BRAGATSTON study is to provide a low cost tool for measuring CAC in breast cancer patients, thereby identifying patients at increased risk of CVD. Breast cancer patients and doctors can act upon this, by adapting the treatment and/or by adopting cardioprotective interventions. Hereby, the burden of CVD in breast cancer survivors can be reduced and better overall survival rates can be achieved.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the second most common cause of death in breast cancer patients. Certain adjuvant treatments (e.g. anthracyclines, radiotherapy) increase the risk of CVD, in particular in patients with pre-existing CVD risk factors. Early identification of these patients enables targeted cardioprotective interventions, and switching to less cardiotoxic treatments. The strongest independent CVD risk factor is the presence and amount of coronary artery calcium (CAC). In clinical practice, CAC is quantified on cardiac CTs. Breast cancer patients treated with radiotherapy routinely undergo planning CTs. These inferior quality CTs may give the opportunity to routinely assess CAC.

The BRAGATSTON study is a multicenter retrospective observational cohort study (UMC Utrecht, Erasmus Medical Center and Radboudumc). The project is divided into three work packages (WP), each WP with a unique aim:

WP 1: To develop/optimize and validate the UMC Utrecht developed automated software to determine the presence and the amount of CAC (CAC score) on radiotherapy planning CT scans of breast cancer patients.

WP 2a: To evaluate the association between CAC score measured automatically on planning CT scans and the risk of incident (non-)fatal cardiovascular events in breast cancer patients.

WP 2b: To evaluate if the association as defined by work package 2a is modified by type of adjuvant treatment.

WP 2c: To evaluate the association between other candidate imaging biomarkers (e.g. calcifications in other structures like the aorta or heart valves, the amount and distribution of body fat, bone characteristics) measured (automatically) on planning CT scans and the risk of incident (non-)fatal (cardiovascular) events in breast cancer patients.

WP 3: To assess the added value of CAC score measured automatically on planning CT scans over classic cardiovascular risk factors and over treatment characteristics to predict (non-)fatal cardiovascular events in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients treated with radiotherapy in UMC Utrecht, Erasmus Medical Center or Radboudumc between 2004-16
* Planning CT scan available
* Age: ≥18 years
* Gender: both genders

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Incident (non-)fatal (cardiovascular) diseases | Up to 13 years of follow-up, in hazard ratios

CONTACTS AND LOCATIONS:
Overall Officials: Helena M. Verkooijen, MD, PhD, Principal Investigator — Imaging Division, University Medical Center Utrecht, Utrecht; Ivana Išgum, PhD, Principal Investigator — Image Sciences Institute, University Medical Center Utrecht, Utrecht; Luca Incrocci, MD, PhD, Principal Investigator — Department of Radiation Oncology, Erasmus Medical Center, Rotterdam; Hanneke Meijer, MD, PhD, Principal Investigator — Department of Radiation Oncology, Radboudumc, Nijmegen
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gal R, van Velzen SGM, Hooning MJ, Emaus MJ, van der Leij F, Gregorowitsch ML, Blezer ELA, Gernaat SAM, Lessmann N, Sattler MGA, Leiner T, de Jong PA, Teske AJ, Verloop J, Penninkhof JJ, Vaartjes I, Meijer H, van Tol-Geerdink JJ, Pignol JP, van den Bongard DHJG, Isgum I, Verkooijen HM. Identification of Risk of Cardiovascular Disease by Automatic Quantification of Coronary Artery Calcifications on Radiotherapy Planning CT Scans in Patients With Breast Cancer. JAMA Oncol. 2021 Jul 1;7(7):1024-1032. doi: 10.1001/jamaoncol.2021.1144. PMID 33956083
- [Derived] Emaus MJ, Isgum I, van Velzen SGM, van den Bongard HJGD, Gernaat SAM, Lessmann N, Sattler MGA, Teske AJ, Penninkhof J, Meijer H, Pignol JP, Verkooijen HM; Bragatston study group. Bragatston study protocol: a multicentre cohort study on automated quantification of cardiovascular calcifications on radiotherapy planning CT scans for cardiovascular risk prediction in patients with breast cancer. BMJ Open. 2019 Jul 27;9(7):e028752. doi: 10.1136/bmjopen-2018-028752. PMID 31352417